CLINICAL TRIAL: NCT03650660
Title: Concordance Between Echocardiographic Assessment Performed in the Initial Phase of Decompensated Cirrhosis With Edema and Ascites by an Expert Intensive Care Physician and a Non-expert Gastroenterologist
Acronym: EchoCirrho
Status: Terminated | Type: Observational
Why Stopped: departure of the principal recruiter in the study
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2017/JFB-01; 2017-A03144-49 (Other: ANSM)
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2020-08

CONDITIONS: Liver Cirrhoses

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with liver cirrhosis
  Interventions: Other: Trans-thoracic ultrasound

INTERVENTIONS:
Other: Trans-thoracic ultrasound — Trans-thoracic ultrasound performed by an expert and a non-expert

SUMMARY:
The investigators hypothesize that trans-thoracic ultrasound performed by non-specialist gastroenterologists with a standard training by intensive care doctors will give equivalent results to those achieved by experts for a simple evaluation of hemodynamic status.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be an adult at least 18 years old
* Patient has known or suspected cirrhosis (diagnosed by biopsy or based on recognized clinical/biological/radiological criteria)
* Admitted to the gastroenterology service for odematous-ascitic decompensation defined by edema of the lower limbs, and/or ascites, anasarca, associated or not with weight gain.

Exclusion Criteria:

* The subject is participating in an interventional study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Patient is pregnant or breastfeeding
* Patient already participated in the study
* Patient with cirrhosis admitted for a different decompensation (active digestive hemorrhage or sepsis)
* Poorly echogenic patient
* Patient withdraws consent
* Patient with anasarca of cardiac origin
* Ultrasound diagnosis of a severe cardiac pathology requiring specialized treatment in intensive care or cardiology (severe cardiac insufficiency, acute pulmonary edema, endocarditis, severe valvulopathy, cardiac tamponade, intracardiac thrombus)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cirrhosis patients admitted to the gastroenterology service for odematous-ascitic decompensation defined by edema of the lower limbs, and/or ascites, anasarca, associated or not with weight gain.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Concordance in Left Ventricular Ejection Fraction measurement on trans-thoracic ultrasound by expert versus a non-specialist gastroenterologist with standard training | 48 hours
  Difference in measured Left Ventricular Ejection Fraction (%)
Concordance in E' wave at the lateral mitral ring and mitral E wave measurement by expert versus a non-specialist gastroenterologist with standard training | 48 hours
  Difference in measured E / E' ratio
Concordance in stroke volume measurement by expert versus a non-specialist gastroenterologist with standard training | 48 hours
  Difference in measured velocity-time integral (cm)

SECONDARY OUTCOMES:
Death rate | Day 28
Duration of hospitalization | End of follow-up (maximum 28 days)
Number of admissions to intensive care | End of follow-up (maximum 28 days)
Consummation of diuretics | Day 0
albumin infusion necessity | Day 0
Use of vasopressors | Day 0
auto ejection fraction measurement on trans-thoracic ultrasound by expert | Day 0
  Doppler
lateral mitral annulus measurement on trans-thoracic ultrasound by expert | Day 0
  Doppler
Mitral E wave measurement on trans-thoracic ultrasound by expert | Day 0
  Doppler
Mitral A wave measurement on trans-thoracic ultrasound by expert | Day 0
  Doppler
Inferior vena cava collapsibility index measurement on trans-thoracic ultrasound by expert | Day 0
  Doppler
Presence of intrapulmonary shunt | Day 0
  Y/N
Presence of aortic stenosis | Day 0
  Y/N
Presence of mitral insufficiency | Day 0
  Y/N
Presence of mitral stenosis | Day 0
  Y/N
left atrium surface area | Day 0
  cm2
left ventricle diameter | Day 0
  mm
Septal wall thickness | Day 0
  mm
Posterior wall thickness | Day 0
  mm
tricuspid annular plane systolic excursion | Day 0
  mm
tricuspid annular plane systolic velocity | Day 0
  cm/s
heart chamber dilation | Day 0
pulmonary arterial hypertension | Day 0
  mmHg
Pericardial effusion | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Jean François Bourgaux, Principal Investigator — CHU Nimes
Locations (1):
- CHU Nimes, Nîmes, France

REFERENCES:
- [Result] Prost A, Bourgaux JF, Louart B, Caillo L, Daurat A, Lefrant JY, Pouderoux P, Muller L, Roger C. Echocardiographic hemodynamic assessment in decompensated cirrhosis: comparison between Intensivists and Gastroenterologists. J Clin Monit Comput. 2023 Oct;37(5):1219-1228. doi: 10.1007/s10877-023-00983-w. Epub 2023 Feb 25. PMID 36840793